CLINICAL TRIAL: NCT02099604
Title: Efficacy and Safety of the Combination Vitamin D (Vit D), With Pegylated Interferon Alpha-2b (PEG-IFN)/Ribavirin (RBV) in Egyptian Patients With Untreated Chronic Hepatitis C: A Phase III Randomized Open-label Clinical Trial
Brief Title: Efficacy and Safety of the Combination Vitamin D With Standard of Care in Egyptian Patients With Untreated Chronic Hepatitis C
Acronym: ViZIR
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study objectives were considered as obsolete regarding the new AAD arrival
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12226 ViZIR
Record Dates: First submitted 2014-03-24; First posted 2014-03-31 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C - Genotype 4; SVR (Sustained Virological Response); Vitamin D; Treatment Naïve
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Vitamin D; Ribavirin; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Experimental): Vitamin D + Pegylated Interferon Alpha 2b + Ribavirin
  Interventions: Drug: Vitamin D + Pegylated Interferon Alpha 2b + Ribavirin
- Standard of Care (No Intervention): Pegylated Interferon Alpha 2b + Ribavirin

INTERVENTIONS:
Drug: Vitamin D + Pegylated Interferon Alpha 2b + Ribavirin — Vitamin D ARM: 28000UI/week during 4 weeks (lead in phase) then 28000 UI/week associated with PegIFN/RBV during 48 weeks
  Other Names: Vidrop; PegIntron; Rebetol
  Arms: Vitamin D

SUMMARY:
The purpose of this study is to show the superiority of a 4 weeks lead-in phase of Vitamin D followed by a 48 weeks combination of Vitamin D with PEG-IFN plus RBV in comparison with standard PEG-IFN + RBV in untreated Egyptian patients with chronic hepatitis C, on the sustained virological response (SVR) at 3 months after end of treatment (week 60).

DETAILED DESCRIPTION:
- Method: Phase III, randomized, open-label superiority clinical trial, among Egyptian patients with chronic hepatitis C.

- Treatment strategy: Vitamin D Arm: Vitamin D over a 4 weeks lead-in phase followed by Vitamin D in combination with PEG-INF plus RBV during 48 weeks. Standard of Care Arm: PEG-INF plus RBV during 48 weeks.

- Main outcome: Proportion of patients with Sustained Virological Response (SVR) as defined by HCV RNA below the detection limit based on quantitative PCR 12 weeks after stopping treatment.

* Sample Size: 520 patients (260 per arm)
* Enrollment period: 12 months
* Patient's participation duration: 62 weeks (SOC Arm), 66 weeks (Vit-D Arm)
* Statistical analysis:

The superiority of the vitamin D arm will be tested against the standard PEG IFN + RBV combination. 260 patients in each arm will give 80% power to document a 12% difference in the SVR rates between the experimental (Vitamin D) and the control (standard treatment) arms..

A futility analysis is planned for this study, in order to be able to interrupt the trial prematurely in case preliminary results show a lack of efficacy of vitamin D.

This analysis will be performed on half of the patients, thus 260 patients (130 patients per arm), on a week 12/14 week criterion (HCV RNA viral load at W12/W14).

ELIGIBILITY:
Inclusion Criteria:

Common with National Program for Viral Hepatitis

* Age: 18 years to 60 years
* Positive HCV antibodies using a third generation test
* Detectable HCV RNA by PCR
* Liver biopsy showing chronic hepatitis with either a METAVIR score F1 with elevated liver enzymes or scores F2/F3
* Naïve to treatment with PEG-IFN and RBV
* HBs antigen negative
* Prothrombin time ≥60 %, normal bilirubin, alpha-foeto protein < 3*normal range of the laboratory, anti-nuclear antibodies<1/160 Effective contraception during the treatment period; no breast-feeding

Specific to the trial

* Prior approval from the Ministry of Health to be treated as part of the National Program with allocation to Peg-IFN α2b treatment
* Living <100 km from Cairo and able to come to the centre every week for the treatment
* Signed informed consent and willingness to participate in the trial
* Naïve to treatment with vitamin D (received vitamin D less than 30 consecutive days in the 3 months preceding inclusion)
* Biopsy slide validated by NHTMRI pathologist

Exclusion Criteria:

Common with National program for Viral Hepatitis

* Serious co-morbid conditions such as severe hypertension, heart failure, significant coronary heart disease, poorly controlled diabetes (HbA1C>8%) , chronic obstructive pulmonary disease
* Major uncontrolled depressive illness
* Solid transplant organ (renal, heart, or lung)
* Untreated thyroid disease
* History of previous anti-HCV therapy
* Body mass index (BMI) greater than 30 kg/m²
* Known human immunodeficiency virus (HIV) coinfection: although HIV testing will not be proposed or done, patients with known HIV coinfection will not be included in the trial
* Anti-HCV therapy contraindications:
* hypersensitivity to one of the two drugs (PEG-IFN, RBV)
* pregnancy or unwilling to comply with adequate contraception
* breast-feeding
* neutropenia (<1500/mm3)
* anaemia (<11g/dL for women ; <12g/dL for men)
* thrombocytopenia (<100,000/mm3)
* elevated creatinin (>1.5mg/dL)
* concomitant liver disease other than hepatitis C (immuno-active chronic hepatitis B, autoimmune hepatitis, alcoholic liver disease, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson disease)
* liver biopsy showing severe steatosis (>66%) and steatohepatitis; decompensated cirrhosis (Child Pugh>A); hepatocellular carcinoma, METAVIR score F4.
* TSH>5 mU/L

Specific to the trial

* Patients allocated to Peg-IFN alpha 2a treatment
* Hypersensitivity to vitamin D
* Vitamin D contraindications:
* hypercalcaemia (fasting calcaemia >105 mg/L or 2.62 mmol/L)
* ratio calciuria / creatininuria (fasting ratio >1 mmol Ca/mmol creatinin)
* hyperphosphatemia (>1.5 mmol/L)
* calcium lithiasis
* patients being treated with thiazide diuretics (risk of hypercalcaemia with vitamin D treatment)
* patients being treated with glucocorticoïds (decrease in vitamin D efficacy)
* postmenopausal women treated by vitamin D and calcium for osteoporosis
* Treatment by vitamin D more than 30 consecutive days in the 3 months preceding inclusion in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Sustained Virological Response (SVR). | 60 Weeks after peg-IFN/RBV initiation
  Proportion of patients with Sustained Virological Response (SVR) as defined by HCV RNA below the detection limit based on quantitative PCR 12 weeks after stopping treatment.

SECONDARY OUTCOMES:
Rapid Virological Response (RVR) | 4 Weeks after peg-IFN/RBV initiation
  HCV RNA at 4 weeks post initiation of combination therapy (PEG IFN + RBV)
Early Virological Response (EVR) | 12 Weeks after peg-IFN/RBV initiation
  HCV RNA at 12 weeks post initiation of combination therapy
End of Treatment Response (ETR) | 48 Weeks after peg-IFN/RBV initiation
  HCV RNA at end of treatment (week 48)
Normalization of ALT during treatment and 12 weeks after the end of treatment | From 2 Weeks after peg-IFN/RBV initiation to End of Follow-up (Week 60)
Incidence of serious adverse events (SAE) grade 3 and 4 (ANRS scale) | From Lead-in phase (Week -4) to End of Follow-up (Week 60)
  incidence of SAE leading to dosage reduction or treatment cessation, percentage of patients treated by EPO and G-CSF
Evolution of FibroScan values between pre-inclusion and week 60 | At Screening Visit 2 (S2) and at End of Follow-up (Week 60)

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Esmat, MD, PhD, Study Chair — NHTMRI, Cairo, Egypt; Arnaud Fontanet, MD, PhD, Study Chair — Institut Pasteur, Paris France
Locations (1):
- NHTMRI, Cairo, Egypt